CLINICAL TRIAL: NCT00531557
Title: Phase IV Cohort Study Assessing Feasibility of Substituting Double Ritonavir-boosted Protease Inhibitors With Ritonavir-boosted Darunavir in HIV-infected Individuals With Viral Suppression on Highly Active Antiretroviral Therapy.
Brief Title: Double Protease Inhibitor to Darunavir Switch Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Dr Mark Nelson, St Stephens Aids Trust
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SSAT022
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: HIV Infections
Keywords: Darunavir; Euglycaemic clamp; HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Darunavir 600mg BID with ritonavir 100mg BID administered orally.
  Interventions: Drug: Darunavir ritonavir

INTERVENTIONS:
Drug: Darunavir ritonavir

SUMMARY:
The purpose of the study is to study the effects of switching from an antiretroviral combination that includes two ritonavir boosted protease inhibitors to replacement of these two protease inhibitors with a new protease inhibitor called Darunavir (also boosted with ritonavir).

The study will investigate the effect of the switch on viral load (the levels of the HIV virus in the blood), on immunological parameters (CD4 count) and on other safety parameters and also on quality of life.

In a subgroup of patients the impact of the switch on the body's response to the hormone insulin will also be measured (Euglycaemic clamp sub group)

DETAILED DESCRIPTION:
HIV-RNA and CD4+ cell count to monitor virological and immunological response on switching to DRV/r.

Routine safety bloods to include haematology and biochemistry (including U&E, fasted glucose and insulin, liver function test, fasting cholesterol and triglycerides and serum lactate measurements).

Quality of life EuroQOL questionnaires at baseline, and throughout the study to evaluate quality of life in the continued treatment/ treatment switch arms.

A sub group of 10 patients will undergo two euglycaemic clamp procedures in order to determine the extent of glucose disposal. The first clamp will be performed prior to the switching from a double boosted PI therapy to DRV/r and the second one following administration of DRV/r for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected as documented by a licensed HIV-1 antibody ELISA test
2. At least 18 years of age
3. Currently on an antiretroviral regimen including a ritonavir boosted double protease inhibitor
4. The subject is virologically suppressed with a viral load < 50 copies/mL for three months or longer
5. The subject has a CD4+ count above 100 cells/mL
6. ≤ Three DRV associated mutations on previous genotypic resistance test -or if no resistance test available, likely to have ≤ four protease inhibitor mutations based on their clinical history
7. If the subject is a woman of child bearing potential, she must agree to use a barrier method of contraception
8. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements

Exclusion Criteria:

1. Pregnant or lactating women
2. Individuals with prior darunavir exposure
3. Previous allergic or hypersensitivity reaction to darunavir
4. Clinical or laboratory evidence of significantly decreased hepatic function or decompensation, irrespective of liver enzyme levels (liver insufficiency)
5. Subjects diagnosed with acute viral hepatitis at screening
6. Subjects with a grade 3 or 4 laboratory abnormality as defined by DAIDS grading table (see appendix 3: DAIDS AE grading Table), with the following exceptions unless clinical assessment foresees an immediate health risk to the subject:

   * Subjects with pre-existing diabetes or with asymptomatic glucose grade 3 or 4 elevations
   * Subjects with asymptomatic triglyceride or cholesterol elevations of grade 3 or 4.
7. Presence of any currently active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV Infection 1993) with the following exceptions: Stable cutaneous Kaposi's Sarcoma (i.e., no internal organ involvement other than oral lesions) that is unlikely to require any form of systemic therapy during the study; Wasting syndrome due to HIV infection.

   Note: An AIDS defining illness that is not clinically stabilized for at least 30 days will be considered as currently active.
8. Active drug abuse, including alcohol or recreational drugs, which, in the opinion of the investigator, is expected to interfere with the subject's ability to adhere to the study procedures and treatment regimen. Subjects on a methadone program will be accepted if deemed appropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects maintaining viral suppression (< 50 copies/mL) | 48 weeks

SECONDARY OUTCOMES:
• CD4+ count at screening, baseline, weeks 4, 12, 24, 36 and at the end of the study period • Viral suppression below 50 copies/mL and below 500 copies/mL at 4, 12, 24, 36 and 48 weeks • Laboratory abnormalities and adverse events at baseline, 4 | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nelson, Principal Investigator — Chelsea & Westminser Healthcare NHS Trust
Locations (1):
- St Stephens Centre, Chelsea & Westminster Hospital, London, United Kingdom